CLINICAL TRIAL: NCT02925078
Title: The Influence of Mucosa Tissue Thickness on Marginal Bone Loss of Implants With Smooth Collars: A Prospective Controlled Trial
Brief Title: Influence of Mucosa Tissue Thickness on Marginal Bone Loss of Implants With Smooth Collars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Professor of Dentistry and Director of Graduate Periodontics, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00095933
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Gingival Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- <2 mm mucosa thickness (Other): A Biohorizons Tapered Internal Implant, Laser-Lok, Resorbable Blast Textured (RBT) will be placed in subjects that have <2 mm mucosa thickness.
  Interventions: Device: Biohorizons Tapered Internal Implant, Laser-Lok, Resorbable Blast Textured (RBT)
- ≥2 mm mucosa thickness (Other): A Biohorizons Tapered Internal Implant, Laser-Lok, Resorbable Blast Textured (RBT) will be placed in subjects that have ≥2 mm mucosa thickness.
  Interventions: Device: Biohorizons Tapered Internal Implant, Laser-Lok, Resorbable Blast Textured (RBT)

INTERVENTIONS:
Device: Biohorizons Tapered Internal Implant, Laser-Lok, Resorbable Blast Textured (RBT) — Placement of implant in a subject with <2 mm mucosa thickness or a subject with ≥2 mm mucosa thickness.

SUMMARY:
The primary objective of this study is to compare the amount of implant marginal bone loss radiographically and probing depth in between thin and thick mucosa group that will receive a machined collar implant.

Null hypothesis is mucosa thickness does not affect implant marginal bone loss on implant with smooth collar.

DETAILED DESCRIPTION:
Twenty eight adult patients who fulfill the inclusion criteria will be divided into 2 groups based upon the mucosa thickness (<2 mm and ≥2 mm). A signed written informed consent will be obtained from all subjects. Subjects will not be screened or treated until an informed consent has been obtained. Patient information will be protected according to the privacy regulations of the federal Health Insurance Portability and Accountability Act of 1996 (HIPAA).

The enrolled patients will receive implants with 1 mm polished collar. Implants will be restored at 4 (±1) months after placement. Outcome analyses will be performed until 1 (±1 month) year after loading and clinical and radiographic parameters will be evaluated to compare clinical outcomes between groups. The primary outcome is implant marginal bone loss and probing depth from clinical and radiographic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Aged ≥18
* In need of one dental implant in the Maxillary or Mandibular area, can be an anterior, premolar, or 1st molar tooth
* Natural adjacent teeth
* Bone height of ≥10mm
* Bone width of ≥5mm
* Good oral hygiene
* Stable periodontium
* Willingness to fulfill all study requirements

Exclusion Criteria:

* Need bone augmentation
* Need one dental implant that is a 2nd or 3rd molar tooth
* Current smoker or quit smoking less than one year
* Pregnant or plan to get pregnant
* Uncontrolled diabetes (HbA1C > 7)
* Medical conditions that may influence the outcome of the study (neurologic or psychiatric disorders, systemic infections )
* Current use of oral bisphosphonates
* History of IV bisphosphonates
* History of radiation therapy in the head and neck area within 4 years
* Poor oral hygiene (plaque score more than 40% based on O'Leary plaque score)
* Once a group has been filled, subjects who meet the criteria of that group will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS MSD PhD, Principal Investigator — Department of Periodontics and Oral Medicine University of Michigan School of Dentistry
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berglundh T, Lindhe J. Dimension of the periimplant mucosa. Biological width revisited. J Clin Periodontol. 1996 Oct;23(10):971-3. doi: 10.1111/j.1600-051x.1996.tb00520.x. PMID 8915028
- [Background] Linkevicius T, Apse P, Grybauskas S, Puisys A. The influence of soft tissue thickness on crestal bone changes around implants: a 1-year prospective controlled clinical trial. Int J Oral Maxillofac Implants. 2009 Jul-Aug;24(4):712-9. PMID 19885413
- [Background] Balshe AA, Assad DA, Eckert SE, Koka S, Weaver AL. A retrospective study of the survival of smooth- and rough-surface dental implants. Int J Oral Maxillofac Implants. 2009 Nov-Dec;24(6):1113-8. PMID 20162117
- [Background] Ochsenbein C, Ross S. A reevaluation of osseous surgery. Dent Clin North Am. 1969 Jan;13(1):87-102. No abstract available. PMID 5249439
- [Background] Anderegg CR, Metzler DG, Nicoll BK. Gingiva thickness in guided tissue regeneration and associated recession at facial furcation defects. J Periodontol. 1995 May;66(5):397-402. doi: 10.1902/jop.1995.66.5.397. PMID 7623260
- [Background] Claffey N, Shanley D. Relationship of gingival thickness and bleeding to loss of probing attachment in shallow sites following nonsurgical periodontal therapy. J Clin Periodontol. 1986 Aug;13(7):654-7. doi: 10.1111/j.1600-051x.1986.tb00861.x. PMID 3531244
- [Background] Abrahamsson I, Berglundh T, Wennstrom J, Lindhe J. The peri-implant hard and soft tissues at different implant systems. A comparative study in the dog. Clin Oral Implants Res. 1996 Sep;7(3):212-9. doi: 10.1034/j.1600-0501.1996.070303.x. PMID 9151585
- [Background] Albrektsson T, Zarb G, Worthington P, Eriksson AR. The long-term efficacy of currently used dental implants: a review and proposed criteria of success. Int J Oral Maxillofac Implants. 1986 Summer;1(1):11-25. No abstract available. PMID 3527955
- [Background] Peri-implant mucositis and peri-implantitis: a current understanding of their diagnoses and clinical implications. J Periodontol. 2013 Apr;84(4):436-43. doi: 10.1902/jop.2013.134001. No abstract available. PMID 23537178
- [Background] Aparna IN, Dhanasekar B, Lingeshwar D, Gupta L. Implant crest module: a review of biomechanical considerations. Indian J Dent Res. 2012 Mar-Apr;23(2):257-63. doi: 10.4103/0970-9290.100437. PMID 22945720
- [Background] Wennerberg A, Albrektsson T, Andersson B. Design and surface characteristics of 13 commercially available oral implant systems. Int J Oral Maxillofac Implants. 1993;8(6):622-33. PMID 8181824
- [Derived] Sabri H, Hazrati P, Tavelli L, Garaicoa-Pazmino C, Calatrava J, Wang HL, Barootchi S. Impact of Peri-Implant Phenotype on Implant Therapy Outcomes: A 5-Year Cohort Analysis on Soft Tissue-Level Implants. J Clin Periodontol. 2025 Dec 12. doi: 10.1111/jcpe.70062. Online ahead of print. PMID 41387987

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | <2 mm Mucosa Thickness | ≥2 mm Mucosa Thickness
Started | 14 | 16
Completed | 13 | 13
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | <2 mm Mucosa Thickness | ≥2 mm Mucosa Thickness | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 4 | 7 | 11
Age, Continuous [Mean (Full Range); unit: years] | 56.54 [36 to 69] | 56.54 [40 to 75] | 56.54 [36 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 8 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Peri-implant Bone Change (Measured in Millimeters) Between Baseline and 12 Months Follow-up.
Description: Radiographic change in remaining bone level (measured in millimeters) between the surgery visit (baseline) and the 12 month follow up visit.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | <2 mm Mucosa Thickness | ≥2 mm Mucosa Thickness
Number analyzed (Participants) | 13 | 13
millimeters | 0.78 (0.66) | 0.61 (0.71)

2. Primary Outcome: Peri-implant Probing Depth Change (Measured in Millimeters) Between Baseline and 12 Months Follow-up.
Description: Change in probing depths (measured in millimeters) around the dental implant between the crown delivery visit and the 12 month follow-up visit.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | <2 mm Mucosa Thickness | ≥2 mm Mucosa Thickness
Number analyzed (Participants) | 13 | 13
millimeters | 0.65 (0.62) | 1.35 (0.58)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during each subject's entire participation in the study (approximately 1.5 years)
Arm/Group | <2 mm Mucosa Thickness | ≥2 mm Mucosa Thickness
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | <2 mm Mucosa Thickness (N=14) | ≥2 mm Mucosa Thickness (N=16)
Hip replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The subject enrolled in the study and at the time did not inform the study team of any need of a hip replacement. 11 months later, the subject told the study team that he had to have his left hip replaced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT02925078/Prot_SAP_000.pdf